CLINICAL TRIAL: NCT01519921
Title: An Open Label Phase IV Multicenter Study for Efficacy and Safety of Peginterferon Alfa-2a (40KD) (PEGASYS®) in Patients With HBeAg Positive Chronic Hepatitis B
Brief Title: A Study of PEGASYS (Peginterferon Alfa-2a (40KD)) in Patients With HBeAg Positive Chronic Hepatitis B.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18495
Record Dates: First submitted 2012-01-05; First posted 2012-01-27 (Estimated); Results first posted 2016-01-25 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-03

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

ARMS (2):
- PEG-IFN alfa-2a (Treatment naïve) (Experimental): Eligible treatment naïve participants received peginterferon alfa-2a (PEGASYS) 180 micrograms (mcg) subcutaneously (SC) once weekly for 48 weeks, followed by 24 weeks of treatment-free follow-up.
  Interventions: Drug: peginterferon alfa-2a [Pegasys]
- PEG-IFN alfa-2a (YMDD mutant) (Experimental): Eligible tyrosine-methionine-aspartate-aspartate (YMDD) mutant participants received PEGASYS 180 mcg SC once weekly for 48 weeks, followed by 24 weeks of treatment-free follow- up. Participants received lamivudine concomitantly for the initial 12 weeks.
  Interventions: Drug: peginterferon alfa-2a [Pegasys]

INTERVENTIONS:
Drug: peginterferon alfa-2a [Pegasys] — Peginterferon alfa-2a (Pegasys) 180 mcg subcutaneously once a week for 48 weeks

SUMMARY:
This study will evaluate the efficacy and safety of PEGASYS (peginterferon alfa-2a) in patients with HBeAg positive chronic hepatitis B. Patients will be stratified into group A (treatment naïve patients) or B (YMDD mutant patients). All patients will receive PEGASYS 180 micrograms subcutaneously once weekly for 48 weeks, followed by 24 weeks of treatment-free follow up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18-65 years of age
* HBsAg +ve for more than 6 months, HBeAg +ve, AntiHBs -ve
* Detectable hepatitis B virus (HBV) DNA (>100,000 copies/mL)

Exclusion Criteria:

* Coinfection with hepatitis A, hepatitis C or human immunodeficiency virus (HIV)
* Evidence of decompensated liver disease
* A medical condition associated with chronic liver disease other than viral hepatitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (3):
- South Korea (3):
  - Busan
  - Daegu
  - Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 150 participants were enrolled in this study conducted from 26 October 2005 to 24 June 2008 at 7 centers in Republic of Korea.
Groups:
- PEG-IFN Alfa-2a (YMDD Mutant): Eligible tyrosine-methionine-aspartate-aspartate (YMDD) mutant participants received PEGASYS 180mcg SC once weekly for 48 weeks, followed by 24 weeks of treatment-free follow- up. Participants received lamivudine concomitantly for the initial 12 weeks.
Period: Overall Study
Arm/Group | PEG-IFN Alfa-2a (Treatment naïve) | PEG-IFN Alfa-2a (YMDD Mutant)
Started | 86 | 64
Completed | 65 | 49
Not Completed | 21 | 15
Not completed — Adverse Event | 10 | 9
Not completed — Lack of Efficacy | 4 | 3
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Treatment refusal | 2 | 1
Not completed — High alanine aminotransferase (ALT) | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were analysed on Intent-to-treat (ITT) population which included all participants who received at least one dose of study drug. The ITT and the safety populations were identical.
Groups:
- PEG-IFN Alfa-2a (Treatment naïve): Eligible treatment naïve participants received PEGASYS 180 mcg SC once weekly for 48 weeks, followed by 24 weeks of treatment-free follow-up.
- PEG-IFN Alfa-2a (YMDD Mutant): Eligible YMDD mutant participants received PEGASYS 180 mcg SC once weekly for 48 weeks, followed by 24 weeks of treatment-free follow- up. Participants received lamivudine concomitantly for the initial 12 weeks.
- Total: Total of all reporting groups
Arm/Group | PEG-IFN Alfa-2a (Treatment naïve) | PEG-IFN Alfa-2a (YMDD Mutant) | Total
Number analyzed (Participants) | 86 | 64 | 150
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.3 (9.20) | 36.8 (9.0) | 35.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 10 | 33
  Male | 63 | 54 | 117

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hepatitis B Virus DNA <100,000 Copies/mL At Week 72
Description: Participants who had Hepatitis B Virus Deoxyribonucleic Acid (HBV-DNA) levels below 100,000 copies per milliliter (mL) at the end of follow-up (EOF) period (24 weeks after the end of treatment) were classified as responders.
Time Frame: Week 72
Population: Intent-to-treat (ITT) population included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PEG-IFN Alfa-2a (Treatment naïve) | PEG-IFN Alfa-2a (YMDD Mutant)
Number analyzed (Participants) | 86 | 64
percentage of participants | 20.9 [12.9 to 31.0] | 21.9 [12.5 to 34.0]

2. Primary Outcome: Percentage of Participants With Hepatitis B Virus e Antigen Loss At Week 72
Description: Participants with loss of hepatitis B virus e antigen (HBeAg) at the EOF period (24 weeks after the end of treatment) were classified as responders.
Time Frame: Week 72
Population: The ITT population included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PEG-IFN Alfa-2a (Treatment naïve) | PEG-IFN Alfa-2a (YMDD Mutant)
Number analyzed (Participants) | 86 | 64
Percentage of participants | 20.9 [12.9 to 31.0] | 23.4 [13.8 to 35.7]

3. Secondary Outcome: Percentage of Participants With ALT Normalization At Week 48 and Week 72
Description: Participants with ALT less than the upper limit of normal (ULN) at end of treatment (EOT) and EOF period were responders.
Time Frame: Week 48 and Week 72
Population: The ITT population included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PEG-IFN Alfa-2a (Treatment naïve) | PEG-IFN Alfa-2a (YMDD Mutant)
Number analyzed (Participants) | 86 | 64
percentage of participants
  Week 48 (EOT) | 34.9 [24.9 to 45.9] | 29.7 [18.9 to 42.4]
  Week 72 (EOF) | 36.0 [26.0 to 47.1] | 29.7 [18.9 to 42.4]

4. Secondary Outcome: Percentage of Participants With Hepatitis B Virus DNA Below the Limit of Detection At Week 48 and Week 72
Description: Participants with HBV-DNA below the limit of detection i.e. <174 copies/mL at EOT and EOF period were responders.
Time Frame: Week 48 and Week 72
Population: The ITT population included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PEG-IFN Alfa-2a (Treatment naïve) | PEG-IFN Alfa-2a (YMDD Mutant)
Number analyzed (Participants) | 86 | 64
Percentage of participants
  Week 48 (EOT) | 10.5 [4.9 to 18.9] | 10.9 [4.5 to 21.2]
  Week 72 (EOF) | 3.5 [0.7 to 9.9] | 9.4 [3.5 to 19.3]

5. Secondary Outcome: Percentage of Participants With a Combined Response At Week 48 and Week 72
Description: A responder with Combined Response was a participant with HBV-DNA<100,000 copies/mL, HBeAg seroconversion (i.e. loss of HBeAg and presence of anti-HBe) and ALT normalization at EOT and EOF period.
Time Frame: Week 48 and Week 72
Population: The ITT population included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PEG-IFN Alfa-2a (Treatment naïve) | PEG-IFN Alfa-2a (YMDD Mutant)
Number analyzed (Participants) | 86 | 64
Percentage of participants
  Week 48 (EOT) | 8.1 [3.3 to 16.1] | 9.4 [3.5 to 19.3]
  Week 72 (EOF) | 9.3 [4.1 to 17.5] | 14.1 [6.6 to 25.0]

6. Secondary Outcome: Percentage of Participants With Hepatitis B Virus e Antigen Seroconversion
Description: A responder was a participant with loss of HBeAg and presence of anti-HBe at EOT and EOF period.
Time Frame: Week 48 and Week 72
Population: The ITT population included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PEG-IFN Alfa-2a (Treatment naïve) | PEG-IFN Alfa-2a (YMDD Mutant)
Number analyzed (Participants) | 86 | 64
Percentage of participants
  Week 48 (EOT) | 15.1 [8.3 to 24.5] | 23.4 [13.8 to 35.7]
  Week 72 (EOF) | 20.9 [12.9 to 31.0] | 21.9 [12.5 to 34.0]

7. Secondary Outcome: Percentage of Participants With Loss of Hepatitis B Surface Antigen At Week 48 and Week 72
Description: A responder was a participant who were analysed with loss of Hepatitis B Surface Antigen (HBsAg) at EOT and EOF period.
Time Frame: Week 48 and Week 72
Population: The ITT population included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PEG-IFN Alfa-2a (Treatment naïve) | PEG-IFN Alfa-2a (YMDD Mutant)
Number analyzed (Participants) | 86 | 64
Percentage of participants
  Week 48 (EOT) | 1.2 [0.03 to 6.3] | 1.6 [0.04 to 8.4]
  Week 72 (EOF) | 1.2 [0.03 to 6.3] | 1.6 [0.04 to 8.4]

8. Secondary Outcome: Percentage of Participants With Hepatitis B Surface Antigen Seroconversion At Week 48 and Week 72
Description: A responder was a participant with loss of HBsAg and presence of anti-HBs at EOT and EOF period.
Time Frame: Week 48 and Week 72
Population: The ITT population included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PEG-IFN Alfa-2a (Treatment naïve) | PEG-IFN Alfa-2a (YMDD Mutant)
Number analyzed (Participants) | 86 | 64
Percentage of participants
  Week 48 (EOT) | 1.2 [0.03 to 6.3] | 0.0 [0.0 to 0.0]
  Week 72 (EOF) | 1.2 [0.03 to 6.3] | 1.6 [0.04 to 8.4]

9. Secondary Outcome: Number of Participants With Any Adverse Events and Any Serious Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence that occurred during the course of the trial after study treatment had started. An adverse event was therefore any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A Serious Adverse Events (SAE) is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect. Participants with any AEs and any SAEs have been presented.
Time Frame: Up to Week 72
Population: Safety population included participants who received at least one dose of study medication and who had at least one post-baseline safety assessment.
Measure: Number; unit: Participants
Arm/Group | PEG-IFN Alfa-2a (Treatment naïve) | PEG-IFN Alfa-2a (YMDD Mutant)
Number analyzed (Participants) | 86 | 64
Participants
  Any AEs | 75 | 54
  Any SAEs | 4 | 5

ADVERSE EVENTS:
Time Frame: Up to Week 72
Description: An AE was defined as any untoward medical occurrence that occurred during the course of the trial after study treatment had started. An AE was therefore any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug.
Groups:
- PEG-IFN Alfa-2a (YMDD Mutant): Group B included tyrosine-methionine-aspartate-aspartate (YMDD) mutant participants who received PEGASYS 180mcg subcutaneously once weekly for 48 weeks, followed by 24 weeks of treatment-free follow- up.
Arm/Group | PEG-IFN Alfa-2a (Treatment naïve) | PEG-IFN Alfa-2a (YMDD Mutant)
Serious Adverse Events (participants affected / at risk) | 4/86 | 5/64
Other Adverse Events (participants affected / at risk) | 69/86 | 52/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-IFN Alfa-2a (Treatment naïve) (N=86) | PEG-IFN Alfa-2a (YMDD Mutant) (N=64)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Appendicitis (Gastrointestinal disorders) | 0 | 1
Exomphalos (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 2
Bronchopneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-IFN Alfa-2a (Treatment naïve) (N=86) | PEG-IFN Alfa-2a (YMDD Mutant) (N=64)
Neutropenia (Blood and lymphatic system disorders) | 21 | 18
Abdominal pain upper (Gastrointestinal disorders) | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 7 | 5
Dyspepsia (Gastrointestinal disorders) | 10 | 1
Asthenia (General disorders) | 7 | 5
Fatigue (General disorders) | 16 | 17
Influenza like illness (General disorders) | 11 | 12
Pain (General disorders) | 13 | 6
Pyrexia (General disorders) | 3 | 6
Liver function test abnormal (Investigations) | 10 | 7
Weight decreased (Investigations) | 5 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 6
Dizziness (Nervous system disorders) | 6 | 2
Headache (Nervous system disorders) | 16 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 10 | 13
Alopecia (Skin and subcutaneous tissue disorders) | 34 | 24
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 12
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 4
Nausea (Gastrointestinal disorders) | 3 | 4
Insomnia (Psychiatric disorders) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.